CLINICAL TRIAL: NCT01145482
Title: Mechanisms of Insulin Facilitation of Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Andreana P. Haley, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2010-05-0007
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Memory Disorders
Keywords: Memory Disorders; Alzheimer's Disease
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease | interventions — Insulin; Insulin Aspart; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin (Experimental): 20 IU of insulin was administered once daily on two occasions in either the first intervention period or second intervention period using a nasal spray bottle
  Interventions: Drug: Insulin
- Saline (Placebo Comparator): 200 micro liters of saline was administered once daily on two separate occasions in either the first intervention period or second intervention period using a nasal spray bottle
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Insulin — 20 IU of insulin was administered once daily on two occasions in either the first intervention period or second intervention period using a nasal spray bottle
  Other Names: NovoLog, 20 IU
  Arms: insulin
Other: Saline — 200 micro liters of saline was administered once daily on two separate occasions in either the first intervention period or second intervention period using a nasal spray bottle
  Other Names: Saline, 200 micro liters
  Arms: Saline

SUMMARY:
The study described in the present application will test the hypothesis that insulin mediated facilitation of memory in Alzheimer's disease (AD) is achieved through enhanced glutamatergic neurotransmission due to improvements in cerebral glucose metabolism. The effect of a single dose of intranasal insulin on memory and cerebral glutamate concentrations in adults with mild AD or amnestic mild cognitive impairment (aMCI), the presumed prodromal phase of AD will be studied. Successful completion of this study may set the stage for a larger-scale treatment trial of intranasal insulin for adults with memory disorders. However, the use of insulin in this manner at this point in time is purely experimental.

DETAILED DESCRIPTION:
The specific aims of this project will be accomplished through a cross sectional repeated measures design in which 15 participants with mild AD or amnestic MCI will undergo assessments of brain structure and function 15 minutes after a single dose of insulin (20 IU) or placebo. Insulin and placebo conditions will be counterbalanced across participants.

Intranasal insulin or placebo administration: Saline and insulin (NovoLog) will be ordered though the UT Student Health Services Pharmacy (Sharon Roberson, Chief Pharmacist) and stored at 4°C, according to standard pharmacy protocols. Three ml doses of saline or insulin will be packaged in nasal spray bottles (e.g., Spectrum Pharmacy Products bottles 969-17404P and actuators 551-24362P) designed to deliver 100μL dose with each spray. A total volume of 200μL will be delivered during each administration (one 100μL dose in each nostril).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable AD
* Age over 21
* Clinical Dementia Rating of 0.5 or 1.0
* Mini Mental State Exam Score>15

Exclusion Criteria:

* preexisting diabetes
* significant neurological disease that might affect cognition, other than AD, including stroke, Parkinson's disease, multiple sclerosis
* severe head injury with loss of consciousness > 30 minutes or with permanent neurological sequelae
* significant medical illness or organ failure, such as uncontrolled hypertension or cardiovascular disease, chronic obstructive pulmonary disease, liver disease, or kidney disease
* current use of anti-psychotic or anti-convulsant medications
* current or previous use of hypoglycemic agents or insulin
* MRI contraindications
* claustrophobia
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreana P Haley, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of texas at Austin, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin First, Then Saline: 20 IU of insulin was administered once daily on two occasions followed by 200 micro liters of saline once daily on two occasions
- Saline First, Then Insulin: 200 micro liters of saline was administered once daily on two occasions followed by 20 IU of insulin once daily on two occasions
Period: First Intervention (1 Day)
Arm/Group | Insulin First, Then Saline | Saline First, Then Insulin
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention (1 Day)
Arm/Group | Insulin First, Then Saline | Saline First, Then Insulin
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Mean age 74.09, SD = 6.54 Gender, Female = 5, Male = 6
Groups:
- Insulin First, Then Saline: 20 IU of insulin was administered once daily on two occasions followed by 200 micro liters of saline administered once daily on two occasions
- Saline First, Then Insulin: 200 micro liters of saline was administered once daily on two occasions followed by 20 IU of insulin administered once daily on two occasions
- Total: Total of all reporting groups
Arm/Group | Insulin First, Then Saline | Saline First, Then Insulin | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (8.58) | 74.33 (5.92) | 74.09 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Glutamate Concentration
Description: Glutamate concentration was expressed as the ratio of glutamate to creatine. This was determined using magnetic resonance spectroscopy (MRS), a magnetic resonance technique that uses the same equipment as magnetic resonance imaging (MRI), but allows researchers to extract information about the concentrations of various neurochemicals of neurobiological significance.
Time Frame: 15 minutes post insulin or placebo administration
Population: per protocol
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Insulin | Saline
Number analyzed (Participants) | 11 | 11
ratio | 1.34 (0.12) | 1.34 (0.17)

2. Secondary Outcome: Memory
Description: Memory performance was assessed using delayed recall (number of units recalled) on the Wechsler Memory Scale (WMS-IV) logical memory (story recall) test. Scores represent a sum of recalled units of two different stories after a 30 minute delay. Total scores range from 0 to 50 (0-25 for each story) with higher scores reflecting better memory performance
Time Frame: 15 minutes post insulin or placebo administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin | Saline
Number analyzed (Participants) | 11 | 11
units on a scale | 6.73 (6.25) | 5.36 (2.69)

ADVERSE EVENTS:
Time Frame: immediately following study visits
Arm/Group | Insulin | Saline
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin (N=11) | Saline (N=11)
nausea and urge to vomit (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No